CLINICAL TRIAL: NCT04639232
Title: Multicenter, Randomized, Double-blind Parallel Group Pilot Study to Evaluate the Effect of Consuming a Combination of Probiotic Strains and a Combination of Plant Extracts and a Probiotic Strain on the Production and Nutritional Composition of Breast Milk
Brief Title: Effect of Consuming a Combination of Probiotic Strains and a Combination of Plant Extracts and a Probiotic Strain on the Production and Nutritional Composition of Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P047
Record Dates: First submitted 2020-10-16; First posted 2020-11-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Milk Expression
Keywords: Breastfeeding; Galactogogue; Plant extracts; Probiotics
MeSH Terms: conditions — Breast Milk Expression; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): Volunteers will take 6 capsules per day for 28 days a capsule containing maltodextrin.
  Interventions: Dietary Supplement: Placebo
- Prob-milk (Experimental): Volunteers will take 6 capsules per day for 28 days a capsule containing the probiotics combination.
  Interventions: Dietary Supplement: Prob-milk
- Voluntas-Prob (Experimental): Volunteers will take 6 capsules per day for 28 days a capsule containing the combination of plant extracts and the inactivated probiotic strain
  Interventions: Dietary Supplement: Voluntas-Prob

INTERVENTIONS:
Dietary Supplement: Placebo — Each participant will consume 6 capsules daily, 2 in every meal, without any restriction in the diet nor in their habits of life.
  Arms: Control group
Dietary Supplement: Prob-milk — Each participant will consume 6 capsules daily, 2 in every meal, without any restriction in the diet nor in their habits of life.
  Arms: Prob-milk
Dietary Supplement: Voluntas-Prob — Each participant will consume 6 capsules daily, 2 in every meal, without any restriction in the diet nor in their habits of life.
  Arms: Voluntas-Prob

SUMMARY:
The objective of this trial is to evaluate the effect of the consumption of a combination of probiotic strains (Prob-milk) and of a combination of plant extracts plus an inactivated probiotic strain (VoluntasProb) on the production volume and the nutritional composition and the microbiota. of breast milk in lactating women.

DETAILED DESCRIPTION:
Previous studies have shown the galactogogue effect of fenugreek, fennel, and milk thistle. However, to date no study has considered the evaluation of all three extracts. Additionally, certain probiotic strains of Lactobacillus and Bifidobacterium also appear to increase milk production in animal studies.

The objective of this trial is to evaluate the effect of the consumption of a combination of probiotic strains (Prob-milk) and of a combination of plant extracts plus an inactivated probiotic strain (VoluntasProb) on the production volume and the nutritional composition and the microbiota. of breast milk in lactating women. This is a preliminary study whose purpose is to gather information for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Lactating women between 18 and 45 years old, who have given birth to a healthy baby at term (born between 37 and 42 weeks).
2. Who have the perception of having little volume of milk or a nutritional composition of milk that is not adequate for their baby
3. That they are between week 2 and week 6 of breastfeeding, and that at the time of beginning the study they are not supplementing with formula milk the feeding of their baby.
4. That they have the firm intention of breastfeeding for 28 more days.
5. Women who agree to participate and have read, understood and signed the informed consent

Exclusion Criteria:

1. Suffering from any disease that may hinder or prevent breastfeeding
2. Being currently consuming or having consumed in the two weeks prior to the study a probiotic or a supplement with plant extracts.
3. Being consuming any drug that can alter the volume or composition of breast milk.
4. Have an allergy to any antibiotics or peanuts
5. Have an allergy to any of the components of the products under study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breastfeeding mothers
Enrollment: 58 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Volume of breast milk | 28 days
  The volume of breast milk production will be measured as the difference in weight in grams of the child before and after the first and last feeding of the day, measured on two consecutive days. It should be collected on the first two days before starting treatment and two days in a row separated by one week during treatment.
Microbiota of breast milk | 28 days
  Load of Lactobacillus, Bifidobacterium, Staphylococcus, Streptococcus in breast milk

SECONDARY OUTCOMES:
Nutritional composition of breast milk | 28 days
  Analysis of the content of proteins, fatty acids profile and total fat content, and iron and calcium content in breast milk
Measurement of IL-8 in breast milk | 28 days
  Analysis of the concentration of IL-8 (pg/mL) in breast milk
Measurement of IgA in breast milk | 28 days
  Analysis of the concentration of IgA (ug/mL) in breast milk
Baby feces microbiota | 28 days
  Presence of Lactobacillus spp, Bifidobacterium spp., Streptococcus spp. Staphylococcus spp, Bacteroides spp, E. coli spp, Clostridium spp in baby faeces
Baby's anthropometric measures_weight | 28 days
  Weight (kg) of the baby at baseline, 14 days and 28 days.
Baby's anthropometric measures_height | 28 days
  Height (cm) of the baby at baseline, 14 days and 28 days.
Baby's anthropometric measures_BMI | 28 days
  BMI (kg/m2) of the baby at baseline, 14 days and 28 days.
Data about the intestinal health of the baby_stool frequency | 28 days
  Data about stool frequency (times per day)
Data about the intestinal health of the baby_color of the faeces | 28 days
  Data about color of the feces (yellow, mustard, brown, grey, or green)
Data about the intestinal health of the baby_consistency of the feces | 28 days
  Data about consistency of the feces (hard lumps, sausage with cracks, soft sausage, mushy (like porridge),or watery)
Data about sleep parameters of the baby | 28 days
  Hours of night sleeping per day and hours of total sleeping during the day
Infantile colick symptoms | 28 days
  Presence of infantile colick defined as vigorous and inconsolable crying for more than 3 hours a day for at least 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Blanco Rojo, PhD, Principal Investigator — Biosearch S.A.
Locations (1):
- Centro de Salud de Maracena, Maracena, Granada, Spain

IPD SHARING:
Plan to Share IPD: No